CLINICAL TRIAL: NCT07288697
Title: Dose-Dependent Effects of Intraoperative Tranexamic Acid on Surgical Bleeding and Transfusion Requirements in Multilevel Thoracolumbar Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Belgüzar Özsert Bilgin, Assistant Doctor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KDrLKSH-AVR-BOB-01
Record Dates: First submitted 2025-12-02; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Spinal Disorders; Degenerative Spine Disease; Blood Loss, Surgical
Keywords: Tranexamic acid; Spinal surgery; Bleeding; Blood transfusion
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose tranexamic acid (Active Comparator): low-dose TXA (n= 31): 5 mg/kg loading + 1 mg/kg/h infusion
  Interventions: Drug: low-dose TXA
- high-dose tranexamic acid (Active Comparator): high-dose TXA (n = 31): 10 mg/kg loading +2 mg/kg/h infusion
  Interventions: Drug: high-dose TXA

INTERVENTIONS:
Drug: low-dose TXA — low-dose TXA (n= 31): 5 mg/kg loading + 1 mg/kg/h infusion
  Other Names: Tranexamic acid loading; Tranexamic acid infusion
  Arms: low-dose tranexamic acid
Drug: high-dose TXA — high-dose TXA (n = 31): 10 mg/kg loading +2 mg/kg/h infusion
  Other Names: Tranexamic asid loading; Tranexamic asid infusion
  Arms: high-dose tranexamic acid

SUMMARY:
Multilevel spinal stabilization surgery is frequently associated with substantial blood loss and increased transfusion requirements. Tranexamic acid (TXA), an antifibrinolytic agent, reduces perioperative bleeding, but the optimal intravenous dosing regimen remains controversial.

This study aimed to compare the efficacy and safety of two TXA dosing protocols in patients undergoing ≥3-level spinal stabilization surgery.

DETAILED DESCRIPTION:
Multilevel spinal stabilization surgery is frequently associated with substantial blood loss and increased transfusion requirements. Tranexamic acid (TXA), an antifibrinolytic agent, reduces perioperative bleeding, but the optimal intravenous dosing regimen remains controversial.

This study aimed to compare the efficacy and safety of two TXA dosing protocols in patients undergoing ≥3-level spinal stabilization surgery.In this prospective, randomized trial, 62 adult patients scheduled for elective thoracolumbar stabilization involving three or more levels were assigned to receive either low-dose TXA (n= 31): 5 mg/kg loading + 1 mg/kg/h infusion or high-dose TXA (n = 31): 10 mg/kg loading +2 mg/kg/h infusion.TXA was administered intravenously 15 minutes before incision.

Intraoperative blood loss, transfusion requirements, perioperative laboratory values, and complications (thromboembolic, neurological, renal, allergic, and seizure-related) were recorded. Patients were monitored for 48 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 years
* Scheduled for elective ≥3-level spinal stabilization surgery under general anesthesia

Exclusion Criteria:

* History of thromboembolic events
* Myocardial infarction
* Stroke
* Hepatic or renal failure,
* Known allergy to TXA
* Bleeding or coagulation disorders,
* ASA physical status IV
* Trauma or tumor surgery
* Refusal to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative Blood Loss [Milliliters] | During the operation
  The total amount of blood lost during surgery, measured in milliliters.
Number of Patients Requiring Intraoperative Erythrocyte Suspension Transfusion [Number of Participants] | During the operation
  Number of participants who required intraoperative erythrocyte suspension (ES) transfusion.

SECONDARY OUTCOMES:
Postoperative Hemoglobin Level at 24 and 48 Hours [g/dL] | 24 and 48 hours postoperatively
  Hemoglobin values measured at 24 and 48 hours after surgery.
Postoperative Hematocrit Level at 24 and 48 Hours [Percent (%)] | 24 and 48 hours postoperatively
  Hematocrit levels measured at 24 and 48 hours after surgery.
Postoperative Platelet Count at 24 and 48 Hours [×10⁹/L or per mm³] | 24 and 48 hours postoperatively
  Platelet count measured at 24 and 48 hours after surgery.
Aspartate Aminotransferase (AST) Level at 24 and 48 Hours [U/L] | 24 and 48 hours postoperatively
  Biochemical Parameters
Alanine Aminotransferase (ALT) Level at 24 and 48 Hours [U/L] | 24 and 48 hours postoperatively
  Biochemical Parameters
Blood Urea Nitrogen (BUN) Level at 24 and 48 Hours [mg/dL] | 24 and 48 hours postoperatively
  Biochemical Parameters
Creatinine Level at 24 and 48 Hours [mg/dL] | 24 and 48 hours postoperatively
  Biochemical Parameters
Incidence of Postoperative Nausea and Vomiting [Number of Participants] | First 48 hours postoperatively
  Number of participants experiencing nausea and vomiting within 48 hours after surgery, potentially related to tranexamic acid (TXA) administration.
Incidence of Serious Adverse Events Related to Tranexamic Acid [Number of Participants] | First 48 hours postoperatively
  Number of participants experiencing serious adverse events attributable to tranexamic acid use.

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr. Lütfi Kırdar Şehir Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No